CLINICAL TRIAL: NCT00486486
Title: A 3-month, 4-centre, Crossover, Double-masked Study Investigating the 24-hour Intraocular Pressure Control With the Bimatoprost/Timolol Fixed Combination Dosed Morning, or Evening in Subjects With Exfoliative Glaucoma
Brief Title: 24-hour Intraocular Pressure (IOP) Control With the Bimatoprost/Timolol Fixed Combination
Acronym: BTFC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, AGP Konstas, Professor in Ophthalmology, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: A3241
Record Dates: First submitted 2007-06-13; First posted 2007-06-14 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Glaucoma
Keywords: 24-hour IOP control
MeSH Terms: conditions — Glaucoma | interventions — Bimatoprost

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bimatoprost/Timolol AM therapy (Active Comparator)
  Interventions: Drug: Drug: bimatoprost/timolol fixed combination AM; Drug: Bimatoprost/timolol fixed combination dosed PM
- Bimatoprost/Timolol PM therapy (Active Comparator)
  Interventions: Drug: Drug: bimatoprost/timolol fixed combination AM; Drug: Bimatoprost/timolol fixed combination dosed PM

INTERVENTIONS:
Drug: Drug: bimatoprost/timolol fixed combination AM — 3-month chronic dosing in the morning
Drug: Bimatoprost/timolol fixed combination dosed PM — Evening dosing of bimatoprost/timolol fixed combination for a period of 3 months

SUMMARY:
The objective of this crossover, randomized, placebo controlled, double-masked study is to compare the short-term (12 weeks) mean 24-hour IOP control and safety of the new fixed combination (bimatoprost/timolol, BTFC) given PM with placebo once in the morning, versus BTFC given AM with placebo once in the evening versus bimatoprost given in the evening in patients with exfoliative glaucoma (XFG).

DETAILED DESCRIPTION:
PRIMARY STUDY OBJECTIVES

* To show that the mean 24-hour IOP control obtained with BTFC (morning or evening) is statistically better to that with bimatoprost monotherapy given once on the evening.
* To demonstrate that the fixed combination will provide a significantly better IOP control in the morning when dosed in the evening.
* To test whether the mean 24-hour IOP control obtained with BTFC given once in the evening may be statistically better to that with BTFC given once in the morning.
* To show whether there will be less 24-hour fluctuation of IOP with the evening dosing of BTFC.

STUDY POPULATION

Consecutive newly-diagnosed, or suitably washed-out patients with exfoliative glaucoma (XFG) who exhibit a mean untreated IOP greater than 25 mm Hg at baseline (10:00).

ELIGIBILITY:
Inclusion Criteria:

* The patient is suffering from XFG (if the patient has bilateral XFG, both eyes will be treated, but the worse eye will be selected for the statistical analysis)
* Patient is older than 39 years and younger than 85 years
* Patient is able and willing to participate in the study for the whole duration of the follow up. Will sign the consent form.
* At screening the untreated IOP at 10:00 (± 1 hr) is greater than 25 mm Hg and lower than 40 mm Hg
* After bimatoprost run-in therapy the treated IOP at 10:00 (± 1 hr) is greater than 19 mm Hg

Ages: 39 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-03; Primary Completion 2008-05 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Mean 24-hour IOP | 3 months of therapy

SECONDARY OUTCOMES:
Side effects with medications | 3 months of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Anastasios Konstas, MD, PhD, Principal Investigator — Head of the Glaucoma Unit
Locations (2):
- Greece (2):
  - Glaucoma Unit, 1st University Department of Ophthalmology, Thessaloniki, Thessaloniki
  - Glaucoma Unit, 1st University Dept of Ophthalmology, Thessaloniki

REFERENCES:
- [Derived] Konstas AG, Hollo G, Mikropoulos D, Tsironi S, Haidich AB, Embeslidis T, Georgiadou I, Irkec M, Melamed S. Twenty-four-hour intraocular pressure control with bimatoprost and the bimatoprost/timolol fixed combination administered in the morning, or evening in exfoliative glaucoma. Br J Ophthalmol. 2010 Feb;94(2):209-13. doi: 10.1136/bjo.2008.155317. Epub 2009 Oct 12. PMID 19825835